CLINICAL TRIAL: NCT05817357
Title: Use of Air Purification Devices in the Homes of Children and Young People to Improve Respiratory Health - a Pilot Study
Brief Title: Use of Air Purifiers to Improve Respiratory Health in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UoL001754
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Installation of air purifier (Rensair Ltd - Rensair Compact) (Experimental): Rensair Compact air purifier unit will be installed in the homes of all children/young people participating in this study for a period of one-year.
  Interventions: Device: Rensair Compact air purifier unit

INTERVENTIONS:
Device: Rensair Compact air purifier unit — Installation of Rensair Compact air purifier (Rensair Ltd.) in the homes of children/young people participating in this study

SUMMARY:
The goal of this pilot study is to investigate if installing an air purifier in the homes of children and young people with asthma improves their asthma outcomes.

The main questions it aims to answer are:

* Does installing an air purifier in the homes of children and young people with asthma improve their asthma outcomes
* Is the use of an air purifier in the home acceptable to children and young people and their families?

Children and young people with asthma attending our clinic will be selected at random to be invited to take part. For those that take part, an air purifier (Rensair Ltd. - Rensair Compact) will be installed in their home for a one-year period. Data will be collected on numbers of asthma attacks, rescue oral steroids, quality of life, symptoms, lung function at the beginning and at three-monthly intervals throughout the study period. The acceptability to children and young people and their families taking part in this study of using an air purifier in their home will also be assessed.

DETAILED DESCRIPTION:
The goal of this pilot study is to investigate if installing an air purifier in the homes of children and young people with asthma improves their asthma outcomes.

The main questions it aims to answer are:

* Does installing an air purifier in the homes of children and young people with asthma improve their asthma outcomes (including reduction in asthma exacerbations, improvement in symptom control, improvement in quality of life).
* Is the use of an air purifier in the home acceptable to children and young people and their families?

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 to 15 years old
* Attend the asthma clinic in our hospital
* Have a confirmed physician-diagnosis of asthma from the asthma clinic
* Live in mainland England (this is due to delivery of the air purification units and also associated maintenance of them)

Exclusion Criteria:

* Nil specific other than not meeting inclusion criteria

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Number of asthma exacerbations (asthma attacks) | 12 months
  Asthma attacks and unscheduled healthcare visits due to acute asthma (including ED attendance, admission, GP/primary care attendance) - assessed by questionnaire and hospital-recorded attendances/admissions
Number of rescue oral steroid courses | 12 months
  Number of rescue oral steroid courses - assessed by questionnaire and prescription data
Quality of life - mini paediatric asthma quality of life questionnaire score | 12 months
  Quality of life using mini paediatric asthma quality of life questionnaire - the higher the score the better the quality of life
Asthma control test score | 12 months
  Asthma control test (ACT) or child asthma control test score (cACT) - depending on age of participant - the higher the score the better the asthma control
Amount of asthma reliever medication use per week | 12 months
  Amount of use of asthma reliever medication use over a one week period (assessed as a categorical value)
Number of school days absent due to asthma | 12 months
  Number of school days missed due to asthma - assessed by questionnaire
Number of parent/carer work days missed due to their child's asthma | 12 months
  Number of work days missed due to child's asthma - assessed by questionnaire
Forced expired volume in one second (FEV1) | 12 months
  Spirometry measurements using ERS/ATS criteria and Global Lung Initiative Reference z-score
Forced vital capacity (FVC) | 12 months
  Spirometry measurements using ERS/ATS criteria and Global Lung Initiative Reference z-score
FEV1:FVC | 12 months
  Spirometry measurements using ERS/ATS criteria and Global Lung Initiative Reference z-score
Measurement of fraction of exhaled nitric oxide (FeNO) | 12 months
  Fraction of exhaled nitric oxide measurements
Acceptability to children and families participating of using an air purifier in their home | 12 months
  Acceptability to children and young people and their families taking part in the study in terms of use of air purifier in their homes - assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: karl A Holden, Principal Investigator — University of Liverpool
Locations (1):
- Alder Hey Children's Hospital, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No